CLINICAL TRIAL: NCT06735859
Title: Impact of Eating Window and Sleep Disorders on Glycemic Control, Cardiovascular Risk, and Weight Loss in Chronic Diseases
Brief Title: Eating Window and Sleep Disorders on Glycemic Control, Cardiovascular Risk, and Weight Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Sao Jose do Rio Preto Medical School (Other)
Responsible Party: Principal Investigator, Luciana Pellegrini Pisani, Impact of Eating Window and Sleep Disorders on Glycemic Control, Cardiovascular Risk, and Weight Loss in Chronic Diseases, Federal University of São Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 82942424.9.1001.5505
Record Dates: First submitted 2024-12-08; First posted 2024-12-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Hypertension; Obesity and Type 2 Diabetes; Cardiovascular Diseases
Keywords: type 2 diabetes; hypertension; obesity; cardiovascular diseases; nutritional intervention; sleep; eating window
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Obesity; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This study is a randomized, crossover clinical trial with a washout period and follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daytime eating window (7 am - 7 pm) (Active Comparator): Participants will be instructed to follow the assigned eating window for a period of 6 months. In the daytime eating window, there will also be encouragement for sleep hygiene practices.
  Interventions: Behavioral: Comparison of eating windows intervention
- Nighttime eating window (12 pm - 12 am) (Active Comparator): Participants will be instructed to follow the assigned eating window for a period of 6 months.
  Interventions: Behavioral: Comparison of eating windows intervention

INTERVENTIONS:
Behavioral: Comparison of eating windows intervention — Participants will be randomized into two groups to follow either a daytime or nighttime eating window, with normocaloric meal plans based on the Mediterranean diet adapted to Brazilian culture. The first intervention phase will last 6 months, followed by a 3-month washout period during which participants return to their usual eating patterns. After the washout, participants will resume the same eating window for an additional 6 months. A final follow-up assessment will be conducted 3 months post-intervention to evaluate the stability of behavioral changes.

SUMMARY:
This project aims to offer a quantitative and qualitative nutritional approach, along with educational nutritional guidelines for participants with Non-Communicable Chronic Diseases. The main goals are: 1- Regularization of eating habits and windows; 2- Modulation of biochemical, anthropometric, and cardiovascular parameters; 3- Increase in knowledge about healthy eating. In this way, participants will undergo a complete nutritional assessment, comprising anthropometry, biochemistry, clinical, and dietary evaluations.

DETAILED DESCRIPTION:
The study will be conducted at the Endocrinology and Hypertension Clinic of the São José do Rio Preto Medical School between 2026 and 2027, with the objective of collecting comprehensive data for an in-depth analysis of the participants. Eligible individuals will be randomly assigned to two intervention groups. Participants in the first group will follow a daytime eating window (7:00 a.m. to 7:00 p.m.), while those in the second group will follow a nighttime eating window (12:00 p.m. to 12:00 a.m.). Nutritional consultations will be conducted individually at five assessment points: Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), and Month 18 (follow-up). Each consultation will last approximately one hour per participant, and all participants will receive appointment reminders via phone or WhatsApp.

ELIGIBILITY:
Inclusion Criteria:

* Age: Adults >18 years < 80 years; Diagnosis of obesity, diabetes, and hypertension; Gender: Male and female; Availability to attend quarterly meetings over a period of 18 months; Sedentary.

Exclusion Criteria:

* Difficulties in responding to the requested instruments; Impediments to regular attendance in data collection; No diagnosis of Obesity, Diabetes, and Hypertension; Use of insulin therapy, Sodium-Glucose Cotransporter-2 (SGLT-2) inhibitors, and Glucagon-Like Peptide-1 (GLP-1) analogs; Chronic Kidney Disease patients; Normal weight or undernourished individuals; Physical exercise practitioners (>150 minutes of exercise/week).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01-21 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Weight (Kg) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  Weight (kg) will be estimated using the Tanita Tetrapolar Bioimpedance Scale with Octaelectrodes BC 601®. Before the consultation, participants will be instructed to attend the meeting wearing light clothing, avoiding heavy meals, fasting from water for 1 hour, and from caffeine for 24 hours prior to the exam. For the measurements, participants will be asked to remove their shoes and empty their bladder. Subsequently, the individual will be asked to step onto the scale. Data will be collected in the morning to mitigate any type of recurring body water fluctuation throughout the day.

SECONDARY OUTCOMES:
Brain and Muscle ARNT-Like 1 (BMAL1) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  Analyzed the expression of the gene that works in partnership with CLOCK to activate circadian cycle-related genes during the study.
Circadian Locomotor Output Cycles Kaput (CLOCK) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  Analyzed the expression of the gene encoding a key circadian regulatory protein (CLOCK) during the study.
Cryptochrome Circadian Regulator 1 (CRY1) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  Analyzed the expression of the gene encoding a key circadian regulatory protein (CRY1) during the study.
Period Circadian Regulator 1 (PER1) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  Analyzed the expression of the gene encoding a key circadian regulatory protein (PER1) during the study.
Ambulatory Blood Pressure Monitoring (ABPM) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  ABPM will be performed with 24-hour monitoring at five study points to assess circadian blood pressure. Data will include daytime/nighttime averages, dipping patterns, variability, and follow-up changes
Medications | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  Medications will be recorded during the nutritional consultation using the anthropometric and clinical evaluation protocols, aiming to mitigate any bias during the intervention.
Physical exercise | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  The presence or absence of physical exercises was evaluated through conventional qualitative measurement/the survey of the presence or absence of active or sedentary individuals. Patients with levels equal to or greater than 5 trainings sessions per week, with a total duration of 250 min/week, were classified as "active (>5 sessions)/moderate (=5 sessions)". Patients with levels equal to 3 trainings sessions per week, with a total duration of 150 min/week, were classified as "light". Individuals below this recommendation (<3 sessions or zero) were considered to be "sedentary".
Hip Index (HI) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  These are statistical corrections of hip circumference, respectively, normalized for height and weight, providing more accurate information regarding the participant's body composition and cardiovascular risk. HI = HC (cm) ∗ Weight (kg) - 0.482 ∗ Height (cm) 0.31
Neck circumference (cm) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  Neck (cm) circumferences will be measured using the 2.0m Sanny® Anthropometric Tape Measure. Neck circumference will be measured by placing the tape around the neck. The ideal neck circumference is up to 37 cm for men and up to 34 cm for women. Measurements below 39.5 cm for men and 36.5 cm for women are considered to indicate a low risk of heart disease or circulatory disorders.
Hip circumference (cm) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  Hip circumference will be measured with the 2.0m Sanny® measure using the widest point of the hip or the midpoint of the buttocks
HDL cholesterol (mg/dL) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  HDL cholesterol will be measured using the Roche cobas c501® equipment. The adequate levels of HDL cholesterol should be higher than 40 mg/dL of blood.
Triglycerides (TG) (mg/dL) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  triglycerides (TG) will be measured using the Roche cobas c501® equipment. As for the values of the triglycerides, values below 130 mg/dL are desired.
Plasma glucose (mg/dL) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  glucose will be analyzed using Siemens® equipment. For the diagnosis of diabetes, two fasting blood glucose measurements ≥ 126 mg/dL after a minimum of 8 hours of fasting or glycated hemoglobin ≥ 6.5% are considered
Body fat percentage (%) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  body fat percentage (%) will be estimated using the Tanita Tetrapolar Bioimpedance Scale with Octaelectrodes BC 601®. Before the consultation, participants will be instructed to attend the meeting wearing light clothing, avoiding heavy meals, fasting from water for 1 hour, and from caffeine for 24 hours prior to the exam. For the measurements, participants will be asked to remove their shoes and empty their bladder. Subsequently, the individual will be asked to step onto the scale. Data will be collected in the morning to mitigate any type of recurring body water fluctuation throughout the day.
Lean mass (kg) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  lean mass (kg) will be estimated using the Tanita Tetrapolar Bioimpedance Scale with Octaelectrodes BC 601®. Before the consultation, participants will be instructed to attend the meeting wearing light clothing, avoiding heavy meals, fasting from water for 1 hour, and from caffeine for 24 hours prior to the exam. For the measurements, participants will be asked to remove their shoes and empty their bladder. Subsequently, the individual will be asked to step onto the scale. Data will be collected in the morning to mitigate any type of recurring body water fluctuation throughout the day.
Sociodemographic assessment: | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  Sociodemographic assessment: Provides general data such as age, sex, socioeconomic level, race, profession, and others. To classify social classes, the following classifications will be considered: Class A (more than 20 minimum wages); Class B (10 to 20 minimum wages); Class C (four to 10 minimum wages); Class D (two to four minimum wages); and Class E (up to two minimum wages)
Dietary assessment (habitual food recall) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  Dietary assessment (habitual food recall): Analyzes the participant's usual intake, allowing for a thorough evaluation in both quantitative and qualitative aspects, and secondarily in performing calculations/estimates, as well as detecting possible deficiencies/excesses
Skipping breakfast | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  The habit of skipping breakfast will be assessed using the metric "yes" or "no." All data mentioned in this session will be evaluated every three months over the 30 months.
Pittsburgh Sleep Quality Index (PSQI) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  The Pittsburgh Sleep Quality Index (PSQI) is an instrument developed at the University of Pittsburgh, used to identify sleep problems and disorders. It consists of 19 items grouped into seven main components related to sleep:
  Subjective sleep quality: Assesses overall satisfaction with sleep quality.
  Sleep latency: Refers to the time required to fall asleep after going to bed.
  Sleep duration: Measures the total amount of sleep during the night.
  Sleep efficiency: Calculates the proportion of time spent in bed to the total time of sleep.
  Sleep disturbances: Investigates the frequency of problems such as apnea, gasping, and nightmares.
  Use of sleep medication: Identifies the use of substances, such as sleeping pills, to aid sleep.
  Daytime dysfunction: Assesses the impact of sleep on daily functionality, including energy levels and fatigue.
  Participants respond to each item based on their experience over the past 30 days, using a scale of 0 to 3.
Blood pressure (BP) (mmHg) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  Blood pressure (BP) values will be measured using the Omron Digital Control® equipment, after five to ten minutes of rest, with three readings on the right arm (RA) and left arm (LA), with a one-minute interval between measurements. For participants with BP values >160/90 mmHg, a five-minute rest period will be conducted before another measurement is taken. For participants with BP values >200/100 mmHg, where the equipment is unable to measure the pressure, the conventional measurement method using the Nylon Premium Black® sphygmomanometer and Solidor CX® Double Black Stethoscope will be used. Individuals with SBP ≥ 140 mmHg and DBP ≥ 90 mmHg will be considered hypertensive [5,6]. Blood pressure and heart rate data will be evaluated every three months over a 30-month period.
Body Shape Index (ABSI) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  The calculation of allometric indices will be performed: Body Shape Index (ABSI). These are statistical corrections of waist and hip circumference, respectively, normalized for height and weight, providing more accurate information regarding the participant's body composition and cardiovascular risk. ABSI=WC/BMI2/3×height1/2.
Waist/hip ratio | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  The waist/hip ratio will also be calculated by dividing the waist circumference (cm) by the hip circumference (cm). Hip circumference will be measured by placing the tape around the widest part of the hip and the midpoint of the buttocks. Desired values are < 0.85 for women and < 0.9 for men, indicating low cardiovascular risk. Values above these limits are classified as high risk for cardiovascular diseases.
Waist circumference (cm) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  Waist (cm) circumference will be measured using the 2.0m Sanny® Anthropometric Tape Measure. Waist circumference will be measured by placing the tape around the midpoint between the last rib and the hip bone. This point will be marked in advance with a specific pen for anthropometry. Desired waist circumference values are below 80 cm for women and 94 cm for men, indicating "low cardiovascular risk." Values of 80 to 87 cm for women and 94 to 101 cm for men indicate "high cardiovascular risk." Values above 88 cm for women and 102 cm for men indicate "very high cardiovascular risk."
BMI (Body Mass Index - Kg/m²) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  BMI will be calculated using the formula weight (kg) divided by height squared (m)², with the following categories: Underweight < 18.5 kg/m²; Normal weight 18.5 - 24.9 kg/m²; Overweight 25.0 - 29.9 kg/m²; Obesity class 1 30.0 - 34.9 kg/m²; Obesity class 2 35.0 - 39.9 kg/m²; Obesity class 3 ≥ 40 kg/m². For participants > 60 years old, the classification is: Underweight ≤ 22 kg/m²; Normal weight > 22.0 < 27.0 kg/m²; Obesity ≥ 27.0 kg/m²
Height (meters) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  Height (meters) will be measured using the Welmy® stadiometer. The participant will be instructed to position themselves with their back against the stadiometer rod, in an upright posture (looking at the horizon and with the chest expanded).
LDL cholesterol (mg/dL) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  LDL cholesterol will be estimated using the Friedewald Equation ([LDL] = (TC - HDL) - (TG/5)). When triglyceride levels are above 400 mg/dL, LDL cholesterol will be calculated using the Roche cobas c501® equipment with Sekisu® reagents [5,6]. Adequate levels of LDL cholesterol in healthy individuals should be below 130 mg/dL of blood, and for those at risk, levels should not exceed 70 mg/dL.
Total cholesterol (TC) (mg/dL) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  Total cholesterol (TC) will be measured using the Roche cobas c501® equipment. The values of total cholesterol considered to be normal should be below 190 mg/dL, slightly high when they are between 200 and 239 mg/dL, and high when they are above 240 mg/dL.
HbA1c (%) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  HbA1c will be analyzed using Siemens® equipment. For the diagnosis of diabetes, two fasting blood glucose measurements ≥ 126 mg/dL after a minimum of 8 hours of fasting or glycated hemoglobin ≥ 6.5% are considered
Insulin (µU/mL) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  Serum insulin levels will be measured using Siemens® immunoassay equipment. Insulin concentration is a key biomarker for evaluating pancreatic β-cell function and insulin resistance. Reference values: fasting insulin in adults typically ranges from 5-15 µU/mL, with slightly broader ranges observed in children and adolescents (2-25 µU/mL). Elevated fasting insulin levels, in combination with glucose measurements, may indicate impaired glucose metabolism and increased risk for type 2 diabetes.
Creatinine Clearance (24-hour urine, mL/min) | 5 assessment points - Month 0 (baseline), Month 6 (end of first intervention phase), Month 9 (end of washout), Month 15 (end of second intervention phase), FOLLOW-UP Month 18.
  Creatinine clearance will be assessed using 24-hour urine collection and serum creatinine levels, calculated to estimate glomerular filtration rate (GFR). This measure provides an important indicator of renal function and metabolic health. Reference values: adult males (<40 years) typically show 107-139 mL/min, while adult females (<40 years) show 87-107 mL/min. Clearance values decline physiologically by approximately 6.5 mL/min per decade of life. Normal 24-hour urine creatinine excretion ranges from 500-2000 mg/day. Reduced clearance values are associated with impaired kidney function and increased cardiovascular risk.

CONTACTS AND LOCATIONS:
Overall Officials: Luciana P Pisani, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo (UNIFESP), Santos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The study data will be collected, managed, and stored using the REDCap 14.0.9 electronic data capture tools hosted at REDCap - FUNFARME/FAMERP and the database of the Federal University of São Paulo (UNIFESP) - Baixada Santista Campus. After scientific publications, the data will be made available to the scientific community upon request to the researchers responsible for the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will only be available 12 months after publication and will be provided upon formal request to the principal researcher, in accordance with the guidelines of non-paid international journal publishers (subscription option).
Access Criteria: After this period, the data will be provided upon formal request to the principal researcher for up to 6 months. A link will be created with direct access to the data, or upon demand and request, the data will be provided directly to the interested researchers.
URL: https://drive.google.com/drive/